CLINICAL TRIAL: NCT05834803
Title: Effects of Percutaneous Transluminal Renal Angioplasty of Atherosclerotic Renal Artery Stenosis in High-Risk Patients - a Danish Nationwide Randomized Sham-Controlled Study.
Brief Title: Effects of Percutaneous Transluminal Renal Angioplasty of Atherosclerotic Renal Artery Stenosis in High-Risk Patients.
Acronym: DAN-PTRAII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Amsterdam UMC (Other); The Novo Nordic Foundation (Other); The Augustinus Foundation, Denmark. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAN-PTRAII
Record Dates: First submitted 2023-04-03; First posted 2023-04-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Renovascular Hypertension; Renovascular Hypertension With Renal Failure; Heart Failure; Renal Artery Stenosis Atherosclerotic; Percutaneous Transluminal Angioplasty
MeSH Terms: conditions — Hypertension, Renovascular; Heart Failure

STUDY DESIGN:
Intervention Model Description: A Danish Nationwide (3-center) Randomized and Sham-Controlled Study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the operator and his team will know whether the patient receives active treatment or sham treatment. The patient will wear a sleep mask and earplugs during the procedure to ensure blinding. Pressure gradient measurements will be performed in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal artery stenting (Active Comparator): Percutaneous transluminal renal angioplasty with stent placement
  Interventions: Procedure: Renal artery stenting
- Sham procedure (Sham Comparator): Sham procedure
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Renal artery stenting — * Optimal medical therapy, including maximally tolerated renin-angiotensin system blockade with either an angiotensin converting enzyme inhibitor or an angiotensin II receptor blocker
  * Diagnostic tests: Catheter-based angiography and measurement of translesional pressure gradients
  * Treatment: Renal artery stenting performed according to the study protocol
  Arms: Renal artery stenting
Procedure: Sham procedure — * Optimal medical therapy, including maximally tolerated renin-angiotensin system blockade with either an angiotensin converting enzyme inhibitor or an angiotensin II receptor blocker
  * Diagnostic tests: Catheter-based angiography and measurement of translesional pressure gradients
  * Treatment: Sham
  Arms: Sham procedure

SUMMARY:
The goal of this clinical trial is to document a beneficial effect of percutaneous transluminal renal angioplasty (PTRA) of atherosclerotic renal artery stenosis in high-risk patients selected according to the criteria used in the DAN-PTRA study. The main questions the trial aims to answer are if renal artery stenting compared with optimal medical treatment alone has beneficial effects on:

* Blood pressure
* Kidney function
* Hospitalizations for heart failure

DETAILED DESCRIPTION:
Even with optimal medical care, patients with renovascular disease have a very high risk of cardiovascular events and an expected poor outcome. One treatment option of atherosclerotic renal artery stenosis is percutaneous transluminal renal angioplasty with stent placement. Renal artery stenting is, however, still a subject of debate as randomized trials have failed to show a benefit of this compared with optimal medical treatment alone. Following the results of the large CORAL trial in 2014, we established the national prospective DAN-PTRA study using strict and well-defined criteria to select patients for renal artery stenting. In this study, we observed a reduction in blood pressure, an improved kidney function, and a decrease in new hospital admissions due to heart failure after renal artery stenting.

The DAN-PTRAII study is a nationwide high-quality randomized, sham-controlled clinical trial in patients with severe renovascular disease due to atherosclerotic renal artery stenosis. Only patients who fulfill the inclusion criteria on optimal medical treatment can enter the study and only the operator and his team will know whether the patients receive renal artery stenting or sham treatment. Participants will be followed closely for 6 months after the treatment to evaluate the effects of renal artery stenting compared with optimal medical treatment alone on blood pressure, kidney function and hospitalizations due to heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. One or more severe atherosclerotic renal artery stenoses defined as a stenosis ≥70% by catheter-based angiography.
2. In addition, at least one of the following high-risk clinical syndromes:

   1. Resistant hypertension with average 24-hour ambulatory systolic blood pressure ≥150 mmHg despite ≥3 antihypertensive drugs including a diuretic, if tolerated, and each prescribed at optimal doses.
   2. Rapidly declining kidney function with a reduction in estimated GFR of >5 mL/min per 1.73m2 per year and average 24-hour ambulatory systolic blood pressure ≥140 mmHg despite ≥3 antihypertensive drugs including a diuretic, if tolerated, and each prescribed at optimal doses.
   3. Hospital admissions with acute decompensated heart failure (≥2 hospitalizations for heart failure or ≥1 hospitalizations for sudden, "flash" pulmonary edema) with no obvious explanations such as nonadherence, left ventricular ejection fraction <40%, or valvular heart disease and average 24-hour ambulatory systolic blood pressure ≥140 mmHg despite ≥3 antihypertensive drugs including a diuretic, if tolerated, and each prescribed at optimal doses.

All 24-hour ambulatory blood pressure monitorings are performed after nurse-administered medication.

Exclusion Criteria:

* Unable to provide informed consent.
* Treatment-resistant heart failure episodes presumed caused by renovascular disease.
* Rapidly declining kidney function/acute kidney failure approaching the need for dialysis presumed caused by renovascular disease.
* Fibromuscular dysplasia or other non-atherosclerotic renal artery stenosis known to be present prior to randomization.
* Pregnancy or unknown pregnancy status in female of childbearing potential.
* Kidney size <7 cm (pole to pole length) supplied by target vessel.
* Previous kidney transplant.
* Previous PTRA treatment.
* Presence of a renal artery stenosis not amenable for treatment with a stent.

Patients who are not eligible for randomization but treated with renal artery stenting outside the protocol are followed according to the DAN-PTRAII protocol in order to account for all PTRA treatments performed in Denmark in the study period.

Patients treated with renal artery stenting without randomization in the study period include patients with:

1. Treatment-resistant heart failure episodes presumed caused by renovascular disease.
2. Rapidly declining kidney function/acute kidney failure approaching the need for dialysis presumed caused by renovascular disease.
3. At least one of the listed high-risk clinical syndromes AND one or more significant atherosclerotic renal artery stenoses defined as a stenosis of 50-69% by catheter-based angiography with:

   * a mean translesional gradient of ≥10 mm Hg, or
   * a systolic translesional gradient of ≥20 mm Hg, or
   * a renal fractional flow reserve (Pd/Pa) of ≤0.8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory systolic blood pressure. | Baseline and 6 months.
  Change in 24-hour ambulatory systolic blood pressure from baseline to 6 months after renal artery stenting compared with optimal medical therapy alone.

SECONDARY OUTCOMES:
Change in kidney function. | Baseline, Day 1, Day 7, Day 21, 6 weeks, 3 months, and 6 months.
  Change in kidney function (estimated glomerular filtration rate) from baseline to 6 months after renal artery stenting compared with optimal medical treatment alone.
Changes in antihypertensive treatment. | Baseline, 3 months, and 6 months.
  Changes in antihypertensive treatment (both defined daily dose [DDD] and number of agents) from baseline to 6 months after renal artery stenting compared with optimal medical treatment alone.
Change in 24-hour ambulatory systolic blood pressure (statistically adjusted for treatment changes). | Baseline, 3 months, and 6 months.
  Change in 24-hour ambulatory systolic blood pressure from baseline to 6 months after renal artery stenting compared with optimal medical therapy alone, with systolic blood pressure values adjusted for changes in the defined daily doses (DDD) of antihypertensive medications. A change of 1 DDD corresponds to a 5 mmHg change in systolic blood pressure.
Number of participants with cardiovascular and kidney outcomes. | From baseline to 6 months after PTRA/sham.
  Clinical events from baseline to 6 months after renal artery stenting compared with optimal medical treatment alone.
  Clinical events are defined using the same criteria as in the Cardiovascular Outcomes in Renal Atherosclerotic Lesions (CORAL) study except for progressive renal insufficiency (in the CORAL study defined as a reduction from baseline of 30% or more in the estimated GFR).
  Clinical events included in the composite endpoint from baseline to 6-month follow-up:
  1. Death from cardiovascular causes
  2. Death from renal causes
  3. Stroke
  4. Myocardial infarction
  5. Hospitalization for congestive heart failure
  6. Progressive renal insufficiency (a reduction from baseline of 50% or more in estimated GFR)
  7. Permanent renal-replacement therapy
  Only the first event per participant is included in the composite.
Number of deaths from any cause. | From baseline to 6 months after PTRA/sham.
  Death from any cause from baseline to 6 months after renal artery stenting compared with optimal medical treatment alone.
Health status on 12-Item Short Form Survey (SF-12). | Baseline, 3 months, and 6 months.
  Changes in 12-item short form health survey (SF-12) from baseline to 6 months after renal artery stenting compared with optimal medical treatment alone.
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Number of serious adverse events (SAEs), procedure-related complications, and postoperative complications. | From baseline to 30 days after PTRA/sham.
  All serious adverse events, procedure-related complications (≤ 24 hours), and postoperative complications (> 24 hours) occurring within 30 days after the procedure will be systematically recorded, including:
  1. Death from any cause
  2. Rupture, dissection, occlusion, or perforation of the renal artery
  3. Stent thrombosis of the PTRA-treated renal artery
  4. Embolic complications affecting the kidney or peripheral circulation (upper or lower extremity depending on access site)
  5. Bleeding requiring transfusion
  6. Embolization or nephrectomy due to bleeding or other complications
  7. Access-related complications requiring treatment: bleeding, thrombosis, or pseudoaneurysm
  8. Need for acute dialysis
  9. Clinical events as defined in item 5
Evaluation of Diagnostic Techniques. | From baseline to 6 months after PTRA/sham.
  As part of the study, the applicability of diagnostic techniques that remain insufficiently described in the context of renal artery stenosis will be evaluated separately according to the protocol. The following examinations will be assessed: (a) Doppler ultrasound, (b) echocardiography, (c) renography, (d) invasive pressure measurements across stenoses, (e) computational fluid dynamics (CFD) simulations, and (f) proteomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Reinhard, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense C

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Horne AL, Dapolite LA. Protocol for pharmacist management of antineoplastic drug-induced adverse effects in outpatients. Am J Health Syst Pharm. 1997 Mar 15;54(6):680-3. doi: 10.1093/ajhp/54.6.680. No abstract available. PMID 9075498